CLINICAL TRIAL: NCT07132476
Title: The Construction and Validation of a Risk Prediction Model for Perioperative Hypoglycemia in Digestive Endoscopy
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: hexiaoyingningbo1
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypoglycemia group
  Interventions: Other: No adjuvant therapy

INTERVENTIONS:
Other: No adjuvant therapy — Observe and record hypoglycemia

SUMMARY:
Digestive endoscopic surgery, including diagnosis and treatment interventions, has become an indispensable means of managing various gastrointestinal diseases in modern gastroenterology practice. Perioperative hypoglycemia is a common but not fully recognized complication. The reported incidence rate of different study populations and types of surgery ranges from 6.75% to 17.50%. The clinical consequences of endoscopic hypoglycemia are profound. Recurrent attacks are associated with an increased risk of transient ischemic attacks and other cardiovascular and cerebrovascular events. From the perspective of the healthcare system, hypoglycemia may reduce patients' compliance with the intake of intestinal cleaning agents, leading to inadequate intestinal preparation, affecting the effectiveness of diagnosis and treatment, prolonging endoscopic surgery time, increasing hospitalization days and costs. This study aims to develop and validate a comprehensive nomogram that integrates three key dimensions: traditional metabolic risk factors (diabetes status, fasting time), program variables (infusion rate, somatostatin use), and new psychosocial factors (anxiety, sleep quality). By using machine learning enhanced logistic regression to prospectively collect data from 610 patients from multiple centers, the resulting column chart model provides clinical doctors with a practical tool for personalized risk stratification and targeted intervention measures, such as reducing anxiety protocols or optimizing fluid management for high-risk patients. The purpose of this study is to identify the influencing factors of hypoglycemia during the perioperative period of digestive endoscopy, help identify and screen high-risk populations, provide theoretical basis for the development of intervention measures, reduce the occurrence of hypoglycemia during the perioperative period of endoscopy, improve patient satisfaction, and reduce hospitalization time and costs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;

  * Endoscopic surgical methods include endoscopic retrograde cholangiopancreatography (ERCP), endoscopic mucosal resection/stripping (endoscopic mucosal resection, EMR/endoscopic submucosal dissection, ESD), high-frequency electroresection or cold resection of polyps, endoscopic hemostasis, and endoscopic ultrasound-guided puncture, etc.; ③ Patients who have given informed consent and voluntarily participate in the survey.

Exclusion Criteria:

① Those who cannot cooperate with the questionnaire survey;

② Those who cannot cooperate with postoperative diet and fluid management or blood glucose monitoring.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endoscopic treatment and surgery
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
hypoglycemia | perioperative period of the endoscopic
hypoglycemia | the perioperative period of the endoscopic

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] He X, Yang Y, Han Y, Zhang Z. Development and validation of a novel nomogram incorporating psychosocial factors for predicting hypoglycemia during perioperative period of digestive endoscopy (DREAM-Hypo Model). BMC Gastroenterol. 2025 Oct 16;25(1):740. doi: 10.1186/s12876-025-04315-x. PMID 41102649